CLINICAL TRIAL: NCT00274378
Title: Allomatrix Injectable Putty in Distal Radius Fractures. Protocol for a Randomised, Controlled Clinical Study in Unstable Fractures of the Distal Radius
Brief Title: Allomatrix Injectable Putty in Distal Radius Fractures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Stryker Trauma and Extremities (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Allomatrix radius UCL
Record Dates: First submitted 2006-01-06; First posted 2006-01-10 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Radius Fractures
Keywords: radius fracture; fracture fixation; homologous bone transplantation
MeSH Terms: conditions — Radius Fractures

INTERVENTIONS:
Device: ALLOMATRIX injectable putty in distal radius fractures

SUMMARY:
Allomatrix is a combination of Demineralized Bone Matrix with a binding medium of calcium sulfate hemihydrate and carboxymethylcellulose. Allomatrix combines the osteoinductive capacity of DBM with the osteoconduction and controlled resorption of surgical grade calcium sulfate.

Unstable fractures of the distal radius do not resist displacement once it has been manipulated into an anatomical position.

There is a parallel between the quality of the anatomic result and the residual capacity of the wrist, except in older, low demanding patients.

Injectable osteoconductive cements have been introduced to fill voids in metaphyseal bone and may provide a better stability around hardware in osteoporotic bone and help maintain reduction of fracture fragments.Moreover, a product like ALLOMATRIX could accelerate and improve bone healing and fracture stability by its osteoinductive properties. However, the clinical significance of these new bone graft materials still have to be proven in a randomised controlled study set-up.

DETAILED DESCRIPTION:
STUDY DESIGN

The study is designed as a randomised, prospective, study with concurrent control. A total of 50 patients will be enrolled by one centre and will be randomised into two groups. One group of patients (comprising 50% of the study population) will have ALLOMATRIX Injectable Putty implanted. In a control group of patients (comprising 50% of the study population as well ) no graft material will be used.

Patients will be randomly assigned to one of the two treatment arms. Sequentially numbered randomisation envelopes will be provided. Once the surgical reduction and stabilisation has been completed, the next sequentially numbered randomisation envelope will be opened and the patient will receive the treatment listed within the envelope. Each envelope will contain one of the treatment arms based on a computer generated randomised schedule.

DURATION AND ENDPOINTS OF THE STUDY The enrollment period is expected to be about 3 years. Patients will be followed from a pre-operative visit through a one-year visit.

Study End Points:

* Comparison of time to healing of the fracture
* Comparison of function of operated wrist
* Radiographic and densitometric assessment of bone regeneration
* Failure rates (Non-union, malunion, fracture instability, wrist stiffness)
* Complication rates (infection, drainage, hardware failure, wound dehiscence)
* Bone growth factors (on blood samples from both forearms at 3 weeks after surgery)

PATIENT SELECTION

The study is directed to unstable distal radius fractures among types I, III and V, according to the classification of Fernandez (4).

It was decided to follow a group of younger patients because the outcome in older, low demand patients is not significantly dependent of a precise reduction contrary to the outcome in younger, high demand patients (15).

STUDY: PRACTICAL INFORMATION

1. For each patient presenting as a candidate for the study, the inclusion and exclusion criteria should be reviewed. After informed consent, pre-operative data are collected (see case report form) and regular pre-operative data are collected to plan the operation. The patient is usually operated within one week after the injury with distal radius fracture.
2. The treatment protocol of distal radius fractures relies on a decision scheme developped by Fernandez and Wolfe (21). We favored percutaneous stabilisation over open reduction and internal fixation. No significant clinical difference was noted between those two techniques in unstable fractures (22). The surgical procedure is conducted under brachial plexus anesthesia.For type I and III (4), the fracture is reduced manually with image intensifier control. One or two Kirshner wires (1.5mm) are directed from the tip of the radial styloid dorsally to the first extensor compartment at an angle of approximately 45 degrees to cross the fracture and enter the dorsoulnar cortex of the radius proximally to the fracture. These wires are placed using a power drill. An additional wire is placed into the fracture fragment, inserted into the dorsoulnar corner of the radius between the fourth and fifth extensor compartments and directed from dorsoulnarly towards palmar radially in a distal to proximal direction.6 The tips of the wires are bent and left just outside the skin, if necessary resorbable sutures (Vicryl 3/0) are used. For type III fractures (4), an external fixator bridging the joint completes usually the procedure. The criteria for reduction3 are an ulnar inclination of 22°, a palmar inclination of 11°, neutral ulnar variance and radial width (distance from the most lateral tip of the radial styloid process to the longitudinal axis through the center of the radius on an AP film). A radioscopic image of the contralateral wrist is taken in the operating room to serve as control, in the same prosupination conditions, to be standardized in the radiology department(19,20). The angles are measured preoperatively with an appropriate software (OEC radioscopy ) and controlled postoperatively with the same radioscopy software.

At the end of the surgical reduction and stabilization of the fracture, the sequentially numbered randomization envelope will be opened and the patient will receive the treatment listed within the envelope : either the ALLOMATRIX Injectable Putty or no additional graft.

ELIGIBILITY:
Inclusion Criteria:

* unstable distal radius fracture

Exclusion Criteria:

* associated traumatic lesions
* associated severe pathological conditions
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Hand ability: self-assesment questionnaire ABILHAND and DASH

SECONDARY OUTCOMES:
Bone mineral density
Radiological evaluation
Hand impairment (strength, sensibilty, mobility)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier BARBIER, MD, Principal Investigator — Cliniques Universitaires St-LUC, 1200 Brussels
Locations (1):
- Cliniques Universitaires St-Luc, Brussels, Belgium

REFERENCES:
- [Background] Cassidy C, Jupiter JB, Cohen M, Delli-Santi M, Fennell C, Leinberry C, Husband J, Ladd A, Seitz WR, Constanz B. Norian SRS cement compared with conventional fixation in distal radial fractures. A randomized study. J Bone Joint Surg Am. 2003 Nov;85(11):2127-37. doi: 10.2106/00004623-200311000-00010. PMID 14630841
- [Background] Barbier O, Penta M, Thonnard JL. Outcome evaluation of the hand and wrist according to the International Classification of Functioning, Disability, and Health. Hand Clin. 2003 Aug;19(3):371-8, vii. doi: 10.1016/s0749-0712(02)00150-6. PMID 12945633
- [Background] Lafontaine M, Hardy D, Delince P. Stability assessment of distal radius fractures. Injury. 1989 Jul;20(4):208-10. doi: 10.1016/0020-1383(89)90113-7. PMID 2592094
- [Background] Hollevoet N, Verdonk R. Outcome of distal radius fractures in relation to bone mineral density. Acta Orthop Belg. 2003 Dec;69(6):510-4. PMID 14748106